CLINICAL TRIAL: NCT04698070
Title: Evaluation of Two Optimizing and Simplifying Strategies on Acute Malnutrition Treatment in Children Aged 6 to 59 Months in Mirriah District, Zinder, Niger
Brief Title: Optimizing Acute Malnutrition Management in Children Aged 6 to 59 Months in Niger (OptIMA Niger)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35237
Record Dates: First submitted 2020-12-19; First posted 2021-01-06 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Acute Malnutrition in Infancy (Disorder)
Keywords: Acute malnutrition; Randomized Clinical Trial; Child Malnutrition; Severe acute malnutrition; Moderate acute malnutrition; Niger; Sub-Saharan Africa; MUAC
MeSH Terms: conditions — Child Nutrition Disorders; Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard (Active Comparator): RUTF 130-200 kcal/kg/day for children with nutritional edema or MUAC < 115 mm or WHZ <-3 and RUSF 500 kcal/d for children 6-23 months with WHZ between -2 and -3 Z and MUAC 115-124 mm.
  Interventions: Other: National nutritional Strategy (Niger)
- OptiMA (Experimental): RUTF 170 kcal/kg/d for children with nutritional edema or MUAC < 115 mm; 125 kcal/kg/d for MUAC 115-119 mm and 75 kcal/kg/d for MUAC 120-124 mm.
  Interventions: Dietary Supplement: Nutritional Strategy - OptiMA
- ComPAS (Experimental): RUTF 1000 kcal/d for children with nutritional edema or MUAC < 115 mm and 500 kcal/day for MUAC 115-124 mm.
  Interventions: Dietary Supplement: Nutritional Strategy - ComPAS

INTERVENTIONS:
Dietary Supplement: Nutritional Strategy - OptiMA — All children randomized to this arm will be treated with a RUTF, with weekly ration determined according to MUAC, weight and presence of nutritional edema. Ration will be adjusted weekly according to the change in MUAC and weight throughout the outpatient follow-up until the child achieves nutritional recovery.
  RUTF dosage will 170 kcal/kg/d for the most severely wasted (MUAC < 115 mm or edema) and reduced to 125 kcal/kg/d for children with MUAC 115-119mm and 75 kcal/kg/d for children with MUAC 120-124 mm.
  All children will be followed-up for 6 months following randomization. They will have weekly outpatient visit in the health facility until they meet nutritional recovery criteria, and then a monthly community-based follow-up in their villages (vital status, anthropometric measures and clinical condition). Referral to the health facility for appropriate nutritional/medical care if illness or acute malnutrition relapse detected).
  Arms: OptiMA
Dietary Supplement: Nutritional Strategy - ComPAS — All children randomized to this arm will be treated with RUTF, with weekly ration determined according to MUAC and presence of nutritional edema. Children enrolled with MUAC < 115 mm or edema will receive 1000 kcal/d (2 sachets/day) RUTF until MUAC has surpassed 115 mm and/or edema is resolved for 2 weeks at which time ration will be reduced to 500 kcal/d (1 sachet/day) until MUAC > or = to 125 mm is achieved for 2 consecutive weeks. Children enrolled with MUAC 115-124 mm will receive 1 sachet/day until MUAC > or = 125 mm is achieved for 2 consecutive weeks and clinically well. Following nutritional recovery, a study nurse will conduct monthly community-based follow-up in their villages (vital status, anthropometric measures and clinical condition) with referral to the health facility for appropriate nutritional/medical care if illness or acute malnutrition relapse detected) for the remainder of the 6 month period following inclusion.
  Arms: ComPAS
Other: National nutritional Strategy (Niger) — Different protocols for SAM and MAM comprise the Niger National Nutrition Protocol:
  1. SAM: Children with MUAC<115 or WHZ<-3 or nutritional edema, will be treated with RUTF, according to a dosage table based on weight at each visit.
  2. MAM: Children aged between 6-24 months with MUAC between 115 -124 mm and WHZ>-3 will be treated with RUSF. Children with the same anthropometry but age 24-59 m will only receive supplementation if they develop criteria for SAM during the 6 month study period. They will be monitored via monthly home visits by a study nurse.
  All children will be followed-up for 6 months following randomization. Children eligible for RUTF at randomization will have a weekly outpatient visit in the health facility until they meet discharge criteria, and then a bi-monthly community-based follow-up in their villages (vital & anthropometric status and referral to the health facility for appropriate nutritional/medical care if indicated).
  Arms: Standard

SUMMARY:
Acute malnutrition (AM) is a continuum condition, arbitrarily divided into severe and moderate categories (SAM, MAM) which are managed separately, with programs overseen by different agencies with different products and supply chains. Such separation complicates delivery of care, contributes to poor program performance, and creates confusion among caregivers. Reduction in the mortality burden from AM will stem from improved simplicity, efficiency and cost-effectiveness of current protocols.

Eligibility for SAM treatment in the current Niger protocol is complex. It is determined by 3 independent criteria: nutritional oedema, Mid-Upper Arm Circumference (MUAC) < 115 mm or weight-height Z score (WHZ) <-3. Also, the Ready to Use Therapeutic Food (RUTF) ration in Niger protocol (130-200 kcal/kg/d) is paradoxical. The amount of RUTF prescribed in the first weeks of treatment is often less than what given to child reaching recovery (MUAC > 125 and WHZ >-2), because weekly ration is determined by the child's weight. Rate of weight gain is highest in the first two weeks of treatment, then plateaus - suggesting no benefit of increased RUTF ration at the end of treatment. Progressive reduction is a more rational use of RUTF and this supplement is equally effective for SAM and MAM.

This community-based non-inferiority trial will compare two strategies for the treatment of AM to the Niger protocol for SAM and MAM. The Optimizing treatment for acute MAlnutrition (OptiMA) strategy uses MUAC < 125 mm or nutritional oedema as admission criteria and optimizes RUTF by adapting doses to the degree of malnutrition. RUTF dose for MUAC < 115 mm or oedema is 170 kcal/kg/d and progressively reduces to 75 kcal/kg/d as MUAC increases. The Combined Protocol for Acute Malnutrition Study (ComPAS) uses the same eligibility criteria like OptiMA, but simplifies more the RUTF ration by providing 1000 kcal/d for children with oedema or MUAC < 115 mm and 500 kg/d for children with MUAC 115-124 mm. Children are considered recovered if they have 2 consecutive weekly MUAC measures ≥ 125 mm.

Children will be individually randomized to treatment in one of the 3 study arms and will attend clinic visits weekly until nutritional recovery. After discharged, they will be monitored monthly via a nurse-conducted home visits until 6 months post-inclusion. The trial arms will be compared using a composite outcome indicator that includes vital status, anthropometric measures and relapse following the index AM episode.

The hypothesis is that simplified strategies could substantially increase the number of children in care compared to current SAM programs without requiring additional RUTF or staffing while maintaining recovery rates in line with current programs.

DETAILED DESCRIPTION:
The main outcome, the success rate, is defined by a composite of three endpoints : alive, not acutely malnourished per the definition applied at inclusion and not having an additional episode of AM throughout the 6- month observation period. All other children are classified as 'unsuccessful'.

The secondary major outcome, the recovery rate, is defined by reaching during the 6 month follow-up a MUAC>=125 and no oedema during two consecutive weeks, a minimum RUTF treatment period of 4 weeks and good clinical condition.

Sample size:

For the main objective, the expected success rate is 68% with a statistical power of 90%. For the secondary priority objective n°1, the expected recovery rate is 82% and for the secondary priority objective n°2, the expected recovery rate is 74% with a statistical power of 80%. For all objectives, the margin of non-inferiority set is 10% with a level of significance set at 1.25% unilaterally. An inflation of 5% to account for unexploitable data was also added. The number of randomized subjects required is:

* 568 participants to meet the main objective;
* 295 participants with severe acute malnutrition to meet the secondary priority objective n°1.
* 384 participants with MUAC<115mm at admission to meet the secondary priority objective n°2.

Data collection and monitoring :

A paper form will be completed by the trial nurses during the outpatient follow-up or at home visits. Data will be recorded by data entry agents supervised by a data manager using RedCAP software.

Data monitoring will be performed every week at each site by clinical trial monitors under the responsibility of the research activities manager, according to the recommendations of Good Clinical Practices. All data entered in the database will be checked for completeness and consistency. The methods of data entry, coding, control, validation and database freezing will be described in a "data management" guide. Before the implementation of the trial, a monitoring plan will be established.

Analysis :

Before the end of the inclusion period, a statistical analysis plan will be established.

The occurrence of the primary endpoint (success rate) will be compared between the OptiMA and ComPAS strategies to the standard protocol.

The occurrence of the primary secondary endpoint (recovery rate) will be compared between the OptiMA and ComPAS strategies to the standard protocol, for children randomized in the severe acute malnourished stratum and for children admitted with a MUAC<115mm.

These comparisons will be made by Intention To Treat (ITT) (including all randomized participants), and Per-Protocol (PP) (including only those participants who received the full randomized treatment strategy).

The primary analysis (success in the overall population regardless of the level of malnutrition) and the main secondary analysis (recovery rate in the "severely malnourished" stratum) in ITT and PP are non-inferiority analyses.

The OptiMA and ComPAS strategies will be deemed non-inferior to the standard strategy if the primary and main secondary analysis statistically demonstrate non-inferiority in both ITT and PP.

The primary analyses in terms of success and recovery will be performed on available data. In case of missing data, a sensitivity analysis will be performed using the maximum bias method. Missing data can be vital status if the child is absent at the last visit, and anthropometric data (weight, MUAC, height). In the case of missing height data, the last available height can be taken into consideration given the low variability of this value from one month to the next.

The probabilities of success, recovery and relapse in each of the strategies and the quantities of RUTF consumed per child to achieve recovery will serve to construct a cost-effectiveness model.

ELIGIBILITY:
Inclusion criteria:

* Age 6 to 59 months old upon study inclusion
* Meet one of the acute malnutrition criteria defined as follows:

  * MUAC < 125mm or
  * Weight for Length Z-score <-3 (WHO standard) or
  * Oedema grade + or ++;
* Resident in health area where the study is conducted ;
* Child's mother or guardian provides informed consent.

Exclusion Criteria:

* Children with medical condition requiring hospitalization or negative appetite test or oedema grade +++;
* Children allergic to milk, peanuts and/or RUTFs ;
* Children diagnosed with a chronic pathology such as sickle cell anemia, trisomy 21, congenital heart disease, neurological condition;
* Children currently enrolled in another malnutrition programme.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2304 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Success rate | 6-month after randomisation
  The primary outcome is a binary composite indicator. Children classified as 'success' fulfil all of the following criteria: alive, not acutely malnourished per the definition applied at inclusion and no additional episode of acute malnutrition (inclusion criteria) throughout the 6-month observation period. All other children are classified unsuccessful.

SECONDARY OUTCOMES:
Recovery rate in children with SAM WHO definition | Throughout the 6-month observation period
  The secondary priority outcome n°1 is the recovery rate in participants with severe acute malnutrition (WHO definition)defined as follows: absence of bipedal oedema and MUAC > 125 mm during two consecutive weeks, a 4-week minimum duration of treatment as clinically well, i.e. axillary temperature <37.5°C. This outcome will be measured throughout the 6-month observation period. All children reaching these criteria during outpatient treatment our during the home visit will be defined recovered.
Recovery rate in children with MUAC<115mm | Throughout the 6-month observation period
  The secondary priority outcome n°2 is the recovery rate in participants with MUAC<115mm defined as follows: absence of bipedal oedema and MUAC > 125 mm during two consecutive weeks, a 4-week minimum duration of treatment as clinically well, i.e. axillary temperature <37.5°C. This outcome will be measured throughout the 6-month observation period. All children reaching these criteria during outpatient treatment our during the home visit will be defined recovered.

OTHER OUTCOMES:
Assess the cost-effectiveness of OptiMA and ComPAS strategies compared to the national protocol of acute malnutrition treatment in Niger | At 6 month
  The ICER (Incremental cost-effectiveness Ratio) will be estimated in each arm.
Outpatient recovery rate | Throughout the 16-weeks outpatient follow up.
  Recovery rate defined as follows: as follows: absence of bipedal oedema and MUAC > 125 mm during two consecutive weeks, a 4-week minimum duration of treatment as clinically well, i.e. axillary temperature <37.5°C will be estimated at the end of the outpatient follow up.
Consumption of RUTF | At the visit of recovery status occuring through the 6 month study completion
  The average number of RUTF sachets per child recovered and per child successfully treated
Recovered children by RUTF quantity | At the visit of recovery status occuring through the 6 month study completion
  The average number of successful and cured children for a given amount of RUTF.
Relapse rate to a new episode of AM and to a new episode of SAM | Throughout the 6-month observation period
  Comparison of the proportion of children who relapse to a new episode of AM and to a new episode of SAM in SAM children at inclusion and in children with AM at inclusion between each arms and risk factors analysis.
Non-response rate | At 16 weeks after inclusion
  Comparison of the proportion of non response (children who did not recovered after 16 weeks under supplementation) in each arms and risk factors analysis.
Recovery rate of children without supplementation | Throughout the 6-month observation period
  Describe the recovery of children not receiving nutritional supplementation with RUTF when included in the standard protocol.
Recovery rate of WaST children | Throughout the 6-month observation period
  Comparison of the recovery rate of children with acute malnutrition associated with severe or moderate stunting in each arms.
Hospitalisation rate | Throughout the 6-month observation period
  Comparaison of the hospitalisation rate in children with AM at inclusion between both arms in each population

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shepherd, MD, Principal Investigator — Alliance for International Medical Action; Renaud Becquet, MPH,PhD,HDR, Principal Investigator — Inserm U1219 Bordeaux Population Health Center
Locations (4):
- Niger (4):
  - Diney, Mirriah, Zinder Region
  - Droum, Mirriah, Zinder Region
  - Gada, Mirriah, Zinder Region
  - Gaffati, Mirriah, Zinder Region

IPD SHARING:
Plan to Share IPD: Yes
The research findings will be disseminated in peer-reviewed journals, meetings and international conferences.
  Individual participant data will be accessible through controlled access repositories, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: SAP : before end of the study on ClinicalTrials.gov Individual participant data : Beginning 6 months and ending 36 months following article publication. After 36 months the data will be available in our University's data warehouse
Access Criteria: Study Protocol and ICF(both in french) can be shared on request Individual participant data : researchers who provide a methodologically sound proposal and whose proposed use of the data has been approved by an independent review committee

REFERENCES:
- [Derived] Daures M, Hien J, Phelan K, Boubacar H, Atte S, Aboubacar M, Aly AAGM, Mayoum B, Azani JC, Koffi JJ, Seri B, Beuscart A, Gabillard D, Hubert V, Cazes C, Kinda M, Anglaret X, Kangas S, Shepherd S, Becquet R. Simplifying and optimising management of acute malnutrition in children aged 6 to 59 months: study protocol for a 3 arms community-based individually randomised controlled trial in decentralised Niger. Trials. 2022 Jan 28;23(1):89. doi: 10.1186/s13063-021-05955-6. PMID 35090531
- See also: Description ALIMA website — http://alima.ngo